CLINICAL TRIAL: NCT04423640
Title: The Analysis of the Inflammatory Response and the Development of Humoral and Cellular Immunity in Patients With Coronavirus Disease 2019 (COVID-19)
Brief Title: Analysis of the Inflammatory Response and the Development of Humoral and Cellular Immunity in Patients With COVID-19
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Coordinación de Investigación en Salud, Mexico (Other Government)
Collaborators: Instituto Mexicano del Seguro Social (Other Government)
Responsible Party: Sponsor
Other Study IDs: R-2020, 3601-043
Record Dates: First submitted 2020-05-27; First posted 2020-06-09 (Actual); Last update posted 2020-08-13 (Actual); Status verified 2020-05

CONDITIONS: SARS-CoV-2

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Whole blood
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- COVID Patients: Diagnosed patients with COVID-19 by PCR
  Interventions: Other: Active COVID-19 disease

INTERVENTIONS:
Other: Active COVID-19 disease — Adult patients admitted to the UMAE Specialty Hospital of CMN SXXI with a diagnosis of COVID-19. The diagnosis must be corroborated by the RT-PCR test.

SUMMARY:
The SARS-CoV-2 infection in the airway epithelium induces cytopathic effects and the cessation of ciliary movement. Increased cytokines and chemokines have been reported to be associated with the severity of the disease. However, most of the molecular and cellular aspects of the inflammatory response and the processes of development of humoral and cellular immunity in these patients are unknown. The aim of this study is characterizing inflammatory processes, seeking to expand the knowledge of the cellular and molecular pathophysiology of COVID-19 that could help in the decision-making of treating health personnel. Mainly, the study is focused on analyzing the inflammatory response by determining cytokines and chemokines. Also, the viral load of the patients with COVID-19 will be determined and will be correlated with the antibody titers. On the other hand, cells will be immunophenotyped to search the cellular depletion profile. Finally, an epidemiological analysis of the patients will be carried out.

ELIGIBILITY:
Inclusion Criteria:

* Patients over 16 years old with positive molecular diagnosis of Covid-19, in the Laboratory of IMSS

Exclusion Criteria:

* Patients with immunosuppressive diseases: HIV +, Hepatitis C virus, primary immunodeficiencies, rheumatoid arthritis, lupus erythematosus and patients under treatment with immunosuppressants

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Mexicans, beneficiaries of the IMSS
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2020-04-15 (Actual); Primary Completion 2020-06-15 (Actual); Study Completion 2020-08-15 (Estimated)

PRIMARY OUTCOMES:
Serum levels of cytokines and chemokines | Day 0
  Pg/ml of IL-2, CXCL8 / IL-8,IL-4, CCL5 / RANTES, IL-6, CXCL9 / MIG, IL-10, CCL2 / MCP-1, TNF-alfa, CXCL10 / IP-10, IFN-alfa, soluble receptor IL6, IFN-gamma.
Serum levels of cytokines and chemokines | Day 3
  Pg/ml of IL-2, CXCL8 / IL-8,IL-4, CCL5 / RANTES, IL-6, CXCL9 / MIG, IL-10, CCL2 / MCP-1, TNF-alfa, CXCL10 / IP-10, IFN-alfa, soluble receptor IL6, IFN-gamma.
Serum levels of cytokines and chemokines | Day 7
  Pg/ml of IL-2, CXCL8 / IL-8,IL-4, CCL5 / RANTES, IL-6, CXCL9 / MIG, IL-10, CCL2 / MCP-1, TNF-alfa, CXCL10 / IP-10, IFN-alfa, soluble receptor IL6, IFN-gamma.
Viral load | Day 0
  log10 U/ml
Viral load | Day 7
  log10 U/ml
Immunophenotype of myeloid cells | Day 0
  Immunophenotypic profile of myeloid cells in COVID by surface molecules CD45, CD14, CD16, mIL-6R, CD73 and CD3. reported in relative fluorescence units and relative percentage of cells analyzed by flow cytometry
Immunophenotype of myeloid cells | Day 3
  Immunophenotypic profile of myeloid cells in COVID by surface molecules CD45, CD14, CD16, mIL-6R, CD73 and CD3. reported in relative fluorescence units and relative percentage of cells analyzed by flow cytometry
Immunophenotype of myeloid cells | Day 7
  Immunophenotypic profile of myeloid cells in COVID by surface molecules CD45, CD14, CD16, mIL-6R, CD73 and CD3. reported in relative fluorescence units and relative percentage of cells analyzed by flow cytometry
RBD-SARS-CoV Protein S- antibodies | Day 0
  relative absorbance units by ELISA
RBD-SARS-CoV Protein S- antibodies | Day 3
  relative absorbance units by ELISA
RBD-SARS-CoV Protein S- antibodies | Day 7
  relative absorbance units by ELISA
Analysis of cellular immune response | Day 0
  Cell count per area (/ mm2) of immune cell sub-populations
Analysis of cellular immune response | Day 3
  Cell count per area (/ mm2) of immune cell sub-populations
Analysis of cellular immune response | Day 7
  Cell count per area (/ mm2) of immune cell sub-populations
Hematopoietic stem cells and progenitor cells populations in peripheral blood | Day 0
  Immunophenotypic profile of stem cells and progenitor cells populations COVID by surface molecules CD34, CD38, CD45RA, Lin, CD3, CD8, CD56, CD19, CD20, CD11b, CD235a andCD14. reported in relative fluorescence units and relative percentage of cells, analyzed by flow cytometry
Hematopoietic stem cells and progenitor cells populations in peripheral blood | Day 3
  Immunophenotypic profile of stem cells and progenitor cells populations COVID by surface molecules CD34, CD38, CD45RA, Lin, CD3, CD8, CD56, CD19, CD20, CD11b, CD235a andCD14. reported in relative fluorescence units and relative percentage of cells, analyzed by flow cytometry
Hematopoietic stem cells and progenitor cells populations in peripheral blood | Day 7
  Immunophenotypic profile of stem cells and progenitor cells populations COVID by surface molecules CD34, CD38, CD45RA, Lin, CD3, CD8, CD56, CD19, CD20, CD11b, CD235a andCD14. reported in relative fluorescence units and relative percentage of cells, analyzed by flow cytometry

SECONDARY OUTCOMES:
Questionnaire of Sociodemographic, labor, pathological and personal characteristics | Day 0
  Questionnaire
SOFA (Secuential Organ Failure Assessment Score) | Day 0
  Is used to track a person's status during the stay in an intensive care unit to determine the extent of a person's organ function or rate of failure. The score is based on six different scores, one each for the respiratory, cardiovascular, hepatic, coagulation, renal and neurological systems.
SOFA (Secuential Organ Failure Assessment Score) | Day 3
  Is used to track a person's status during the stay in an intensive care unit to determine the extent of a person's organ function or rate of failure. The score is based on six different scores, one each for the respiratory, cardiovascular, hepatic, coagulation, renal and neurological systems.
SOFA (Secuential Organ Failure Assessment Score) | Day 7
  Is used to track a person's status during the stay in an intensive care unit to determine the extent of a person's organ function or rate of failure. The score is based on six different scores, one each for the respiratory, cardiovascular, hepatic, coagulation, renal and neurological systems.
Fibrinogen | Day 0
  mg/dL
Fibrinogen | Day 3
  mg/dL
Fibrinogen | Day 7
  mg/dL
C-Reactive protein | Day 0
  mg/L
C-Reactive protein | Day 3
  mg/L
C-Reactive protein | Day 7
  mg/L

CONTACTS AND LOCATIONS:
Overall Officials: Constantino López Macías, PhD, Study Chair — UIMIQ Hospital de especialidades, CMN S.XXI
Locations (1):
- UMAE Hospital de Especialidades del Centro Médico Nacional Siglo XXI, IMSS., Mexico City, Mexico City, Mexico

IPD SHARING:
Plan to Share IPD: Yes
Data of outcomes for meta-analysis purposes
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: After publication for 6 months
Access Criteria: Data for meta-analysis purposes, the review requests will be done by the responsible of the research.